CLINICAL TRIAL: NCT06623097
Title: Exercise and Nutrition for Older Cancer Survivors and Their Support Person: The Vitality Study
Acronym: VITALITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-697
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cancer Survivorship
Keywords: Cancer Survivorship

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Virtually Supervised Care Comparator (Experimental): * Complete virtually supervised exercise sessions 3x weekly with their study partner.
  * Complete Mediterranean eating program coaching session 1x weekly.
  Interventions: Behavioral: Supervised Exercise and Diet Program
- Arm 2: Unsupervised Care (Experimental): * Receives exercise and diet intervention recommendations including 3x weekly workouts and healthy eating goals
  * Weekly recorded informative videos
  * 4x weekly supportive text messages
  * Study website access and interventional booklet
  Interventions: Behavioral: Unsupervised Exercise and Diet Program

INTERVENTIONS:
Behavioral: Supervised Exercise and Diet Program — A home-based, virtually supervised, moderate-to-vigorous aerobic and resistance exercise intervention with a certified cancer exercise trainer. The exercise sessions will include aerobic exercise on a stationary bicycle and total-body resistance training using resistance bands. Stationary bicycle, resistance bands, activity tracking watch, and Wi-Fi enabled tablet (if needed) will be provided to participants. Dyads will receive remotely delivered nutrition coaching sessions (via telephone or video conferencing) with a health coach each week. Mediterranean eating pattern goals will be tracked using the journal feature of the My Wellness Research platform website.
  Arms: Arm 1: Virtually Supervised Care Comparator
Behavioral: Unsupervised Exercise and Diet Program — A home-based, unsupervised moderate-to-vigorous aerobic and resistance exercise intervention. The exercise sessions will include aerobic exercise on a stationary bicycle and total-body resistance training using resistance bands. Stationary bicycle, resistance bands, activity tracking watch will be provided to participants. Dyads will receive Mediterranean eating pattern goals, with an introductory session conducted by research staff. Diet intake will be tracked using the journal feature My Wellness Research platform website.
  Arms: Arm 2: Unsupervised Care

SUMMARY:
This research study will compare the impact of virtually supervised and unsupervised home-based exercise and diet programs on cognitive and physical function among cancer survivors and support persons. This study will involve a 6-month home-based virtually supervised or unsupervised exercise and diet intervention.

The names of the study interventions involved in this study are:

* Virtually supervised exercise and healthy diet care
* Unsupervised exercise and healthy diet care

DETAILED DESCRIPTION:
This is a multi-center, parallel arm, comparative effectiveness trial to compare the impact of supervised and unsupervised home-based exercise and diet programs on cognitive function and physical function among cancer survivors and support persons.

Participants and support persons in this study will be randomly assigned to one of two groups: Group A: Virtually Supervised Care or Group B: Unsupervised Care. Randomization means a participant is placed into a study group by chance.

The research study procedures include screening for eligibility, in-clinic visits, evaluations of fitness, physical health, diet, and cognitive function, surveys, and questionnaires.

Participation in this study is expected to last 36 months.

It is expected about 1528 people will participate in this research study.

Patient Centered Outcomes Research Institute (PCORI) is supporting this research study by providing funding for the study.

ELIGIBILITY:
Inclusion Criteria for Survivor Participants:

* Ability to understand and the willingness to sign informed consent prior to any study- related procedures.
* Older adults (≥65 years of age); cancer survivors who are at higher risk for developing comorbid conditions related to physical and cognitive function due to age declines.
* Completed chemotherapy and/or targeted therapy in the previous 36 months; said treatment exposure negatively impacts cognitive and physical function.
* Diagnosed with breast, lung, prostate, or colorectal cancer which are obesity-related cancers with higher risk for developing comorbid conditions related to physical and cognitive function.
* No detection of dementia as measured by scoring ≥ 23/41 on the Telephone Interview for Cognitive Status (TICS); it may be unsafe for individuals with dementia to participate in the intervention, and they may not be able to experience measurable cognitive improvement. Additionally, scores on cognitive measures could reflect task comprehension failure - not actual cognitive ability - as individuals with dementia may not be able to comprehend or follow the test instructions
* Overweight/obese: BMI ≥25 kg/m2 (calculated using height and weight) or body fat >35% for people assigned female at birth and >25% for people assigned male at birth (estimated by bioelectrical impedance); higher body weight negatively impacts cognitive and physical function.
* Currently participating in <60 minutes of structured moderate-to-vigorous exercise per week (determined by screening questionnaire); sedentary cancer survivors have a higher need and are more likely to benefit from exercise exposure.
* No history of disordered eating; to avoid triggering of past eating disorders with a diet intervention program.
* Reside with an (≥18 years of age) informal support person willing to participate; survivor/support person dyads will participate in the trial together per the goals of the trial and finding mechanism.
* Speak English or Spanish; the study teams will only be able to accommodate for these two languages at this time.
* Willing to travel to the respective site for necessary data collection.

Inclusion Criteria for Support Person:

* Adults ≥18 years of age; the intervention is not designed for adolescent and pediatric populations.
* No detection of dementia as measured by scoring ≥ 23/41 on the Telephone Interview for Cognitive Status (TICS); it may be unsafe for individuals with dementia to participate in the intervention, and they may not be able to experience measurable cognitive improvement. Additionally, scores on cognitive measures could reflect task comprehension failure - not actual cognitive ability - as individuals with dementia may not be able to comprehend or follow the test instructions
* No history of disordered eating; to avoid triggering of past eating disorders with a diet intervention program.
* Speak English or Spanish; the study teams will only be able to accommodate for these two languages at this time.

Exclusion Criteria for Survivor Participants:

* Adult cancer survivors less than 65 years of age.
* Survivors with a TICS score ≤ 22/41
* Survivors with a BMI <25 kg/m2 and body fat <35% for people assigned female at birth and <25% for people assigned male at birth.
* Survivors currently consuming a Mediterranean Diet or meeting 2 or more out of the following 3 Mediterranean eating pattern goals in the prior 6 weeks: ≥3 servings of vegetables per day, ≥ 3 servings of beans and legumes per week, or ≥ 1 serving of nuts per day.
* Survivors with unstable comorbidities that prevent participation in moderate-to-vigorous intensity exercise. Persons with unstable comorbidities may develop unexpected adverse events from exercise. For the purpose of participant safety, as well as because this study involves remote, home-based exercise where close supervision is not possible, participants with unstable medical conditions will be excluded. This will be evaluated through the PAR- Q.
* Subjects with severe psychiatric conditions such as Active Major Depression, Bipolar Disorder, significant Suicidal ideation, and an active substance use and/or substance abuse disorder; these conditions can 1) adversely affect important cognitive test measures and 2) the ability to complete certain circumscribed interventions in the study.
* Subjects who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Survivors receiving treatment for an active malignancy (exceptions are treatment for basal cell carcinoma. They may receive long term treatments for their diagnosed breast, lung, prostate or colorectal cancer including hormone therapy). This study is exclusively targeting survivors post-primary cancer treatment.

Exclusion Criteria for Support Person:

* Support persons less than 18 years of age.
* Support persons with a TICS score ≤ 22/41
* Given the age range of support persons include those in childbearing years, people who are pregnant, or plan to become pregnant during study duration will be excluded due to the unknown nature of exercise on developing fetuses.
* Support persons with unstable comorbidities that prevent participation in moderate-to- vigorous intensity exercise. Persons with unstable comorbidities may develop unexpected adverse events from exercise. For the purpose of participant safety, as well as because this study involves remote, home-based exercise where close supervision is not possible, participants with unstable medical conditions are excluded.
* Support persons with severe psychiatric conditions such as Active Major Depression, Bipolar Disorder, significant Suicidal ideation, and an active substance use and/or substance abuse disorder; these conditions can 1) adversely affect important cognitive test measures and 2) the ability to complete certain circumscribed interventions in the study.
* Support persons receiving treatment for an active malignancy or are less than 10 years from the completion of any cancer treatment (exceptions are treatment for basal cell carcinoma). This is to preserve the "role" of the cancer survivor in the dyad.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1528 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Global Cognition | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  The Montreal Cognitive Assessment (MOCA) will also be used to assess global cognition.
Change in Cognitive Function | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  Cognitive function will be measured using the National Institutes of Health (NIH) toolbox (www.nihtoolbox.org). Within the NIH toolbox, executive function, immediate recall, memory, attention, working memory, and processing speed will be measured.
Change in Physical Function (6-minute walk test) | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  The 6-minute walk test is also conducted to assess aerobic endurance and capacity. Distance achieved during the 6-minute walk test is recorded in meters.
Change Physical Function (Short Physical Performance Battery [SPPB]) | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  The SPPB is comprised of three sections: 1) balance with feet together, semi tandem, and full tandem is held for up to 10 seconds with no support (seconds); 2) usual gait speed over four meters is timed (seconds); and 3) chair stand where the time(s) to complete five chair sit-to-stands is recorded.
Change in Physical Function (Timed-Up-And-Go (TUG) Test) | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  The TUG test times how fast it takes a participant to stand up from a chair, walk around a cone placed three meters away from a chair where they start, and end in a seated position (seconds).
Change in Physical Function (Gait Speed) | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  Gait speed is assessed over a six-meter course with a flat surface, where the time to walk the 15 foot course at a usual and fast pace is recorded (seconds).
Change in Physical Function (Sit-to-Stand Test) | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  The sit-to-stand test involves participants completing as many sit-to-stands from a seated chair position to a standing position with full hip extension in 30 seconds.
Change in Physical Function (Grip Strength) | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  Grip strength is assessed using a hand-held dynamometer on the participant's dominant hand.
Change in Physical Function (Frailty) | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  Overall frailty will be assessed using the Rockwood model, a 42-item questionnaire, and the Fried model, a 5-item questionnaire.
Change in Physical Function (Cardiorespiratory Fitness) | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  Cardiorespiratory fitness will be assessed as VO2peak by a graded maximal bicycle exercise stress test.
Change in Physical Function (Muscular Strength) | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  Muscular strength will be assessed using 1-Repetition Maximum (RM) and will be estimated from 10-RM muscular strength tests.

SECONDARY OUTCOMES:
Accelerometer-Captured Physical Activity | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  Physical activity will be recorded for a week with ActiGraph accelerometer sensor. Physical activity also will be measured by self-report using the modified Godin Leisure-Time Exercise Questionnaire (GLTEQ), a 3-item measure with a score range of less than 14 units to 24 units or more. The higher the weekly total score represents the greater a participant's physical activity. The GLTEQ assesses current participation in any structured exercise and asks the participant how much time they spend exercising in a typical 7-day period.
Patient-Reported Outcome: PROMIS-29 Quality of Life Questionnaire | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  Assessed by the PROMIS-29 Profile v2.0 Questionnaire, a 29-item measure graded on a 5 point Likert scale with answers ranging from 5 (without difficulty/never/not at all) to 1 (unable to do/always/very much) with a total score range of 29 to 140 points. A higher score reflects better quality of life.
Patient-Report Outcome: PROMIS Cognitive Function Questionnaire | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  Assessed by the PROMIS- Cognitive Function - Short Form 4a, a 4-item measure graded on a 5-point Likert scale with answers ranging from 5 (never) to 1 (very often) for a total score range of 4 to 20 points. A higher score reflects better cognitive function.
Mediterranean Eating Pattern | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  A trained health coach will conduct virtual or telephone-based dietary recalls of a non-consecutive weekday and weekend day using the NCI-developed Automated Self-Administered 24-hour (ASA24) recall dietary assessment web-based tool. Calorie intake and nutrient density will be averaged over the two days for each time point.
Alternate Mediterranean Diet Score (aMED) | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  The Alternate Mediterranean Diet Score (aMED) will be calculate by comparing an individual's diet to a traditional Mediterranean eating pattern. The total score for the aMED ranges from 0-9, with a higher score indicating greater adherence to aMED dietary pattern.
Carotenoid Scan | From baseline (month 0) to month 6 (post-intervention) to month 12 (follow-up)
  The Carotenoid Scan will be assessed by a reflection spectroscopy device, Veggie Meter®, to noninvasively assess dermal carotenoids as a biomarker of fruit and vegetable intake. Participants will be instructed to take 3 readings (20 seconds per reading), and an average score will be taken.20 Scores range from 0-800, and higher are associated with fruit and vegetable intake in diverse samples of adults.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu